CLINICAL TRIAL: NCT05315492
Title: Strengthening Addiction Care Continuum Through Community Consortium in Vietnam
Brief Title: Strengthening Community Addiction Services in Vietnam
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Li Li, Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Vietnam Addiction Care
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Addiction, Opioid
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention communes (Experimental): CCC intervention
  Interventions: Behavioral: Community Care Consortium (CCC)
- Control communes (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Community Care Consortium (CCC) — The intervention will train community health workers to take an active role in the drug control and addiction service delivery in the community.
  Arms: Intervention communes

SUMMARY:
This study aims to develop and test an intervention to enhance the addiction service continuum with the joint effort of commune health workers and family members of people who use drugs in Vietnam.

DETAILED DESCRIPTION:
The study will develop and test an intervention to strengthen a continuum of addiction services. The intervention, entitled "Community Care Consortium (CCC)," features community health workers' joint effort with family members to provide patient-centered, individualized addiction care and support. The intervention will be developed and tested through three phases in three regions of Vietnam (Ninh Binh, Da Nang, and Can Tho).

In Phase 1, we will conduct formative studies with commune (community) health workers (CHW), community representatives, PWUD, and their family members to identify barriers to addiction service utilization and discuss potential strategies to establish a continuum of addiction services. Based on the formative study findings, the CCC Intervention and its implementation plans will be developed through workgroup meetings with researchers, community members, and target users.

In Phase 2, the CCC Intervention will be piloted in three communes and revised based on acceptability/feasibility data, process evaluation, and feedback from field staff and participants.

In Phase 3, a randomized controlled trial of the CCC Intervention will be conducted in 60 communes, which will be randomized to either an intervention condition or a control condition (30 communes in each condition). A total of 720 PWUD, 720 of their family members, and 180 commune health workers (CHW) will participate in the study. The intervention outcomes on PWUD, CHW, and family members will be assessed with the data collected at baseline, 3-, 6-, 9- and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Having a history of drug use
* Having disclosed drug using status to at least one of his/her family members and is willing to invite this family member to our study
* Currently residing in the selected communes
* Voluntary written informed consent

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1620 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
PWUD's STTR fulfillment score | Changes from baseline to 3-, 6-, 9- and 12- month follow-ups
  This overall score consists of individual indicators in 4 domains: Seek,Test, Treat, Retain

SECONDARY OUTCOMES:
CHW's addiction-related service provision and support | Changes from baseline to 3-, 6-, 9- and 12- month follow-ups
  CHW's service provision and support such as patient referrals and support for treatment retention measured by frequencies of appointment reminder, follow-up activities

OTHER OUTCOMES:
Family members' support in the 4 domains:Seek,Test, Treat, Retain | Changes from baseline to 3-, 6-, 9- and 12- month follow-ups
  Family member's emotional, informational, monetary support, logistic assistance for PWUD treatment and retention as well as scale measures in their caregiver burden and coping.

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- Vietnam (2):
  - National Institute of Hygiene and Epidemiology, Hanoi
  - Community Health Centers, Ninh Bình

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li L, Nguyen TA, Liang LJ, Lin C, Pham TH, Nguyen HTT, Kha S. Strengthening Addiction Care Continuum Through Community Consortium in Vietnam: Protocol for a Cluster-Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 22;12:e44219. doi: 10.2196/44219. PMID 36947125